CLINICAL TRIAL: NCT06598540
Title: Comparison of Two Nutrition-Based Interventions on Physician Well-being - A Randomized Controlled Trial
Brief Title: Comparison of Two Nutrition-Based Interventions on Physician Well-being
Acronym: COMPASSION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maryam S Makowski, PhD, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 75576
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Self-Compassion; Self-care; Self-care Agency; Self-kindness; Self-valuation
Keywords: self-compassion; physician well-being; diet; diet quality; self-care; physician burnout; self-valuation

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized controlled trial to compare the impact on physician well-being outcomes of a brief mindset intervention that frames daily food choices as an opportunity for demonstrating self-kindness to a brief nutrition education intervention among physicians on burnout, self-compassion, self-kindness, diet quality, and readiness to change in physician during 6-weeks. Surveys will be completed at baseline and in weeks 3 and 6.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants would not know the difference between the two arms of the study other than there are two different behavioral nutrition interventions. The biostatistician analyzing the data would not know which arm of the study participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kindness-focused intervention arm (Experimental): Mindset intervention framing food choices as an opportunity to practice self-kindness. Individuals randomized to this arm will participate in a 15-20-minute live virtual educational session delivered via the Stanford Zoom platform. The recording of the session will be available for 7 days on a private and secure educational platform for those who cannot attend the live session and for future review. After participating in the initial educational session, participants can engage in brief (less than 10 minutes) web-based activities on their own time during weeks 2 and 5.
  Interventions: Behavioral: Kindness-focused
- Health-focused intervention arm (Active Comparator): Brief education intervention framing food choices as a component of a healthy lifestyle. Individuals randomized to this arm will participate in a 15-20-minute live virtual educational session. The recording of the session will be available for 7 days on a private and secure educational platform for those who cannot attend the live session and for future review. After participating in the initial educational session, participants will have the option to engage in brief (less than 10-minute) web-based activities on their own time during weeks 2 and 5.
  Interventions: Behavioral: Health-focused

INTERVENTIONS:
Behavioral: Kindness-focused — This mindset intervention frames food choices as an opportunity to practice self-kindness. Individuals randomized to this arm will participate in a 15-20-minute live virtual educational session delivered via the Stanford Zoom platform. The recording of the session will be available for 7 days on a private and secure educational web-based platform. After participating in the initial educational session, participants will have the option to engage in brief (less than 10-minute) web-based activities on their own time during weeks 2 and 5. Examples of such activities include sharing their experiences about considering food choices as an act of self-kindness with other study participants or writing an encouraging letter to a study participant and physician colleague through the private and secure message board of a web-based educational platform.
  Arms: Kindness-focused intervention arm
Behavioral: Health-focused — Brief education intervention framing food choices as a component of a healthy lifestyle. Individuals randomized to this arm will participate in a 15-20-minute live virtual educational session. The recording of the session will be available for 7 days on a private and secure educational web-based platform. After participating in the initial educational session, participants will have the option to engage in brief (less than 10-minute) web-based activities on their own time during weeks 2 and 5. Examples of such activities include writing a brief statement about their perspective on the usefulness of healthy eating and sharing it with physician colleagues in their group through the private and secure message board of a web-based educational platform.
  Arms: Health-focused intervention arm

SUMMARY:
Several studies have shown that self-valuation (also known as self-compassion) strongly predicts burnout in physicians. Although effective, existing self-compassion cultivation programs designed for physicians have significant time commitments and, historically, have had low physician participation rates. With occupational burnout among US physicians at an all-time high, there is a compelling and urgent need to identify pragmatic approaches to address low levels of self-valuation in physicians. This study aims to test the impact of a brief mindset intervention that frames daily food choices as an opportunity to demonstrate self-kindness on self-valuation and burnout in physicians over 6 weeks. Instilling a mindset shift that enables physicians to practice self-valuation as part of their existing, daily routine amidst extreme time pressures is a pragmatic and potentially powerful vehicle to promote self-valuation for physicians.

DETAILED DESCRIPTION:
We will conduct a randomized controlled trial to compare the impact on physician well-being outcomes of a brief mindset intervention that frames daily food choices as an opportunity for demonstrating self-kindness to a brief nutrition education intervention among physicians. Surveys will be completed at baseline and in weeks 3 and 6 after the start of the intervention.

If this proof-of-concept intervention is effective, it will not only provide evidence regarding the value of the specific intervention tested for increasing self-valuation in physicians but also provide a novel framework for future interventions evaluating the ability of mindset interventions to foster self-valuation and clinician well-being.

Primary outcome measures: percentage change in mean scores from baseline at week 6 in scores of the measures below.

1) Self-valuation: We will use two standardized measures to assess self-valuation:

1a. The 4-item Clinician Self-valuation Scale assesses deferment of self-care to meet work demands and harsh responses to personal imperfections and errors during the past two weeks. (1) This assessment will be collected at baseline, week 3, and week 6.

1b. The 3-item self-kindness subscale of the Modified State Self-Compassion Measure, a validated construct developed by Kristin Neff, PhD in 2021 (2). This assessment will be collected at baseline, week 3, and week 6.

2) We will also evaluate participants' self-reported readiness to practice self-valuation, and the importance and confidence in practicing it on a sliding scale.

3) Burnout: We will use the burnout sub-scales of the validated Stanford Professional Fulfillment Index which includes 4 items evaluating the Work Exhaustion domain of burnout and 6 items assessing the Interpersonal Disengagement domain of burnout over the past 2 weeks. These assessments will be collected at baseline, week 3, and week 6.(3)

Secondary outcome measure: percentage change in mean score from baseline at week 6 in scores of diet quality assessed by the validated 9-item Mini-EAT dietary questionnaire designed to assess diet quality in clinician practice. (4) This assessment will be collected at baseline, week 3, and week 6.

In the final survey ( week 6) we will collect participant feedback about satisfaction with the program and recommendations for improvement.

References:

1. Trockel MT, Hamidi MS, Menon NK, et al. Self-valuation: Attending to the Most Important Instrument in the Practice of Medicine. Mayo Clin Proc. 2019;94(10):2022-2031.
2. Neff, K. D., Tóth-Király, I., Knox, M. C., Kuchar, A., & Davidson, O. (2021). The Development and Validation of the State Self-Compassion Scale (Long-and Short Form). Mindfulness, 12(1), 121-140.
3. Trockel M, Bohman B, Lesure E, et al. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018;42(1):11-24.
4. Lara-Breitinger KM, Medina Inojosa JR, Li Z, et al. Validation of a Brief Dietary Questionnaire for Use in Clinical Practice: Mini-EAT (Eating Assessment Tool). J Am Heart Assoc. 2023;12(1):e025064.

ELIGIBILITY:
Inclusion Criteria:

* Physicians of all genders and racial/ethnic backgrounds licensed to practice medicine in the US, and
* Physicians who spend at least 8 hours per week doing clinical work (based on self-report)

Exclusion Criteria:

* Anyone who is not a licensed physician in the US
* Physicians who are not licensed to practice medicine in the US, and
* Physicians who spend less than 8 hours per week doing clinical work.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Percentage change in mean score of self-kindness from baseline at week 6 | 6 weeks
  The 3-item self-kindness subscale of the Modified State Self-Compassion Measures: A validated construct developed by Kristin Neff, PhD in 2021. This assessment will be collected at baseline, week 3, and week 6. Instructions ask respondents to answer questions about their relevant experience "during the past 2 weeks." An example of an item is "I'm being kind to myself."; Scale items are scored on a 5-point Likert scale (Not at all true for me=1;Very true for me=5).
  The scale range is standardized to 0 to 10. Higher scores are more favorable.
Percentage change in mean score of self-valuation from baseline at week 6 | 6 weeks
  The 4-item Clinician Self-valuation Scale assesses deferment of self-care to meet work demands and harsh responses to personal imperfections and errors during the past two weeks. This assessment will be collected at baseline, week 3, and week 6. Instructions ask respondents to answer questions about their relevant experience "during the past 2 weeks." Example items are "When I made a mistake, I felt more self-condemnation than self-encouragement to learn from the experience" and "I put off taking care of my own health due to time pressure." Scale items are scored on a 5-point Likert scale (always = 0; never = 4) and reverse scored such that higher scores are more favorable. The scale range is 0 to 10.
Changes in Stage of Change from baseline at week 6 | 6 weeks
  Perceptions of importance and confidence in practicing self-valuation will be measured on a sliding scale that ranges from 0 to 10 with higher scores being more favorable. Together, indicate how ready the client is to change target behaviors. Lower scores of both ( less than 30) indicate pre-contemplation stage and higher scores ( more than 90) indicate the maintenance stage in terms of four stages of the change: Precontemplation, Contemplation, Action, and Maintenance. We will also evaluate participants' self-reported readiness (5 option Likert scale from not ready to practice: 0, to have been practicing it consistently for 6 months: 4).These assessments will be collected at baseline, week 3 and week 6.
Physician Burnout | 6 weeks
  We will use the burnout sub-scales of the validated Stanford Professional Fulfillment Index which includes 4 items evaluating the Work Exhaustion domain of burnout and 6 items assessing the Interpersonal Disengagement domain of burnout over the past 2 weeks. This includes 4 items that assess work exhaustion and 6 items that assess interpersonal disengagement. Items are scored on a 5-point Likert scale from "not at all" to "extremely." The average item score from the 10 work exhaustion items and interpersonal disengagement items is used to derive an overall burnout score ranging from 0 to 10 with lower scores being favorable. This assessment will be collected at baseline, week 3 and week 6.

SECONDARY OUTCOMES:
Percentage change in mean scores from baseline at week 6 in diet quality | 6 weeks
  Diet quality: assessed by the validated 9-item Mini-EAT dietary questionnaire designed to assess diet quality in clinician practice. This assessment will be collected at baseline, week 3, and week 6. The scores range from 53 to 72 with scores of less than 61: Unheathy, 61-69: Intermediate, mand ore than 69: Healthy indicating diet qualities respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Makowski, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Because the information in this study is collected from practicing physicians in the US, we want to keep the information confidential and will not be sharing individual participant data.

REFERENCES:
- [Result] Lara-Breitinger KM, Medina Inojosa JR, Li Z, Kunzova S, Lerman A, Kopecky SL, Lopez-Jimenez F. Validation of a Brief Dietary Questionnaire for Use in Clinical Practice: Mini-EAT (Eating Assessment Tool). J Am Heart Assoc. 2023 Jan 3;12(1):e025064. doi: 10.1161/JAHA.121.025064. Epub 2022 Dec 30. PMID 36583423
- [Result] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Result] Neff, K.D., Tóth-Király, I., Knox, M.C. et al. The Development and Validation of the State Self-Compassion Scale (Long- and Short Form). Mindfulness 12, 121-140 (2021). https://doi.org/10.1007/s12671-020-01505-4
- [Result] Trockel MT, Hamidi MS, Menon NK, Rowe SG, Dudley JC, Stewart MT, Geisler CZ, Bohman BD, Shanafelt TD. Self-valuation: Attending to the Most Important Instrument in the Practice of Medicine. Mayo Clin Proc. 2019 Oct;94(10):2022-2031. doi: 10.1016/j.mayocp.2019.04.040. Epub 2019 Sep 19. PMID 31543254